CLINICAL TRIAL: NCT01520675
Title: Endoscopic Versus Surgical Treatment of Chronic Pancreatitis - A Randomized Controlled Trial
Brief Title: Endoscopic Versus Surgical Treatment of Chronic Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pramod Kumar Garg, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IESC/T-187/2010
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; randomized controlled trial; endoscopic therapy; surgery; ESWL
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Active Comparator): Patients will be randomized to surgery
  Interventions: Procedure: surgery
- Endotherapy (Active Comparator): Patients will be randomized to endoscopic therapy
  Interventions: Procedure: Endoscopic therapy

INTERVENTIONS:
Procedure: surgery — Drainage procedure
  Other Names: lateral pancreaticojejunostomy
  Arms: Surgery
Procedure: Endoscopic therapy — pancreatic sphincterotomy, removal of calculi, stenting, ESWL
  Other Names: Pancreatic endotherapy
  Arms: Endotherapy

SUMMARY:
Chronic pancreatitis is a progressive inflammatory disease of the pancreas characterized by destruction of pancreatic parenchyma and subsequent fibrosis. Patients with chronic pancreatitis can be treated with medical management, endoscopic therapy and surgical treatment. Among the various theories of causation of pain in chronic pancreatitis, there is theory of ductal hypertension. In this the pancreatic duct obstruction resulting in ductal dilatation, ductal hypertension and parenchymal hypertension is thought to be the cause of pain. For patients with dilated ducts, ductal decompression is advocated. Ductal decompression can be achieved by endoscopy and by surgery. Surgery comprises of lateral pancreaticojejunostomy with or without headcoring. Endoscopic treatment includes sphincterotomy, dilatation of strictures, removal of stones with or without extracorporeal shock wave lithotripsy (ESWL) and stenting. The pros and cons of endoscopic versus surgical therapy are debated. Lateral pancreaticojejunostomy relieves chronic abdominal pain in 65%-93% of patients. Morbidity and mortality rates are generally low, averaging 20% and 2%, respectively. Long-term follow-up of patients after lateral pancreaticojejunostomy reveals that up to 50% of patients develop recurrent symptoms and 10%-35% fail to obtain pain relief. Studies indicate that more than 60% of patients undergoing pancreatic endotherapy are pain free 1 year after the procedure. There are only two randomized controlled trials comparing endoscopic treatment with the surgical therapy. In this study the investigators will be conducting a randomized trial, to compare endoscopic and surgical treatment of chronic pancreatitis. Outcome variables measured in the study will include pain relief, quality of life, morbidity, mortality, length of hospital stay and changes in pancreatic function.

DETAILED DESCRIPTION:
Chronic pancreatitis is a progressive inflammatory disease of the pancreas characterized by destruction of pancreatic parenchyma and subsequent fibrosis. The prevalence of chronic pancreatitis has been found to be very high in southern India (114-200/100 000 population). Alcohol is the most common etiology worldwide, while idiopathic pancreatitis is the most common type in India and China, accounting for approximately 70% of all cases of chronic pancreatitis. It is a cause of considerable morbidity in the form of pain, steatorrhea and diabetes mellitus. Natural history of chronic pancreatitis is characterized by variable course stretching over decades with recurrent acute pancreatitis in the early stage and steatorrhea, diabetes and pancreatic calcification in the later stages. Pain is a prominent clinical feature of chronic pancreatitis and the most troublesome symptom for which medical attention is often sought. Unfortunately, despite much work, the pathophysiology of pain in CP remains poorly understood. Multiple factors have been suspected, which include inflammation, encasement of sensory nerves by the fibrotic process and neuropathy, and duct obstruction, which can lead to high back pressure and parenchymal ischemia. Increased pressure in the main pancreatic duct is likely to be an important cause of pain, particularly in patients with duct dilatation. This explanation forms the conceptual basis for both endoscopic and surgical drainage procedures. Approximately one half of patients with pain owing to chronic pancreatitis come to an intervention aimed principally at pain relief, along with relief of bile duct, duodenal, and major venous obstruction. Patients with chronic pancreatitis can be treated with medical management, endoscopic therapy and surgical treatment. For patients with dilated ducts, ductal decompression is advocated. The pros and cons of endoscopic versus surgical therapy are debated.

The modified Puestow or lateral pancreaticojejunostomy is the most commonly employed surgical procedure. Lateral pancreaticojejunostomy relieves chronic abdominal pain in 65%-93% of patients. Morbidity and mortality rates are generally low, averaging 20% and 2%, respectively. Long-term follow-up of patients after lateral pancreaticojejunostomy reveals that up to 50% of patients develop recurrent symptoms and 10%-35% fail to obtain pain relief.

Overall more than 60% of patients undergoing pancreatic endotherapy are pain free 1 year after the procedure. There are only two randomized controlled trials comparing endoscopic treatment with the surgical therapy.

Dite et al. reported the first trial. Surgery consisted of resection (80 %) and drainage (20 %) procedures, while endotherapy included sphincterotomy and stenting (52 %) and/or stone removal (23 %). In the entire group, the initial success rates were similar for both groups, but at the 5-year follow-up, complete absence of pain was more frequent after surgery (37 % vs. 14 %), with the rate of partial relief being similar (49 % vs. 51 %). In the randomized subgroup, results were similar (pain absence 34 % after surgery vs. 15 % after endotherapy, relief 52 % after surgery vs. 46 % after endotherapy). The increase in body weight was also greater by 20 - 25 % in the surgical group, while new-onset diabetes developed with similar frequency in both groups (34 - 43 %), again with no differences between the results for the whole group and the randomized subgroup. The authors concluded that surgery is superior to endotherapy for long-term pain reduction in patients with painful obstructive chronic pancreatitis.

Cahen et al. reported the second trial. All symptomatic patients with chronic pancreatitis and a distal obstruction of the pancreatic duct but without an inflammatory mass were eligible for the study. Thirty-nine patients underwent randomization: 19 to endoscopic treatment (16 of whom underwent lithotripsy) and 20 to operative pancreaticojejunostomy. During the 24 months of follow-up, patients who underwent surgery, as compared with those who were treated endoscopically, had lower Izbicki pain scores (25 vs. 51, P<0.001) and better physical health summary scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey questionnaire (P=0.003). At the end of follow-up, complete or partial pain relief was achieved in 32% of patients assigned to endoscopic drainage as compared with 75% of patients assigned to surgical drainage (P=0.007). Rates of complications, length of hospital stay, and changes in pancreatic function were similar in the two treatment groups, but patients receiving endoscopic treatment required more procedures than did patients in the surgery group (a median of eight vs. three, P<0.001). Authors concluded that surgical drainage of the pancreatic duct was more effective than endoscopic treatment in patients with obstruction of the pancreatic duct due to chronic pancreatitis.

Both these trials had a small sample size. The population studied was also different. ESWL was not included in protocol in one of the trials. In one of the trials only pancreatic duct drainage was chosen as the surgical therapy. The proposed study will compare surgery with endoscopic therapy in Indian population with chronic pancreatitis. The outcomes compared would include pain relief, quality of life, morbidity, mortality, length of hospital stay and changes in pancreatic endocrine and exocrine function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis
* Failed medical treatment
* Dilated pancreatic duct ( > 5mm)

Exclusion Criteria:

* Age under 12 or more than 70 years
* Pregnancy
* Multiple (> 3) large stone (> 1.5 cm) in head of pancreas or stones present throughout head, body and tail
* Contraindications to surgery

  * American Society of Anesthesiologists class IV
  * Portal hypertension
* Contraindications to endoscopic treatment

  * Gastrectomy with Billroth II reconstruction
  * Other pancreatitis-related complications requiring surgery
* Previous interventional therapy for chronic pancreatitis

  * Pancreatic endotherapy
  * Previous surgery
* Suspected pancreatic cancer
* Refusal to participate

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 1 year
  Relief in pain

SECONDARY OUTCOMES:
Quality of life | 6 Month
  QoL score
Morbidity | 30 days
  Any comoplications
Mortality | 30 day
  Mortality
Changes in pancreatic endocrine function | 6 Month
  Development or change in diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Agrawal, MS, Principal Investigator — All India Institute of Medical Sciences; T K Chattopadhyay, Study Director — All India Institute of Medical Sciences; Peush Sahni, Study Director — All India Institute of Medical Sciences; Sujoy Pal, Study Chair — All India Institute of Medical Sciences; N R Dash, Study Chair — All India Institute of Medical Sciences; Pramod Garg, Study Director — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India